CLINICAL TRIAL: NCT06696677
Title: Small Intestine Length Measurement Using 3D CT Volumetry and in Vivo Measurement Using Pre-marked Graspers in Revisional Bariatric Surgeries. A Comparative Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsalam M, Associate Professor of General Surgery, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: TSBL06052024
Record Dates: First submitted 2024-10-05; First posted 2024-11-20 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Small Intestine Length
Keywords: Small bowel Length; reconstructed 3D CT scan; Revisions bariatric Surgery

STUDY DESIGN:
Intervention Model Description: This is a prospective cross-sectional analytic study designed to compare two methods of small bowel length measurement: preoperative 3D CT volumetry and intraoperative laparoscopic measurement using pre-marked graspers. The study will include adult patients undergoing revisional bariatric surgeries at Kasr AlAiny Hospitals. All participants will undergo preoperative imaging and intraoperative measurements, with results analyzed to determine the accuracy and correlation between the two methods.
Who Masked: Investigator
Masking Description: the investigator- the surgeon- will not be aware of the pre-operative measurements found in the CT scan, not to be biased in measuring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Marked Laparoscopic graspers group (Active Comparator): in this arm, the graspers will be marked by a sterile tape, 5 cm in length. This will help for accurate measuring of the whole intestine.
  Interventions: Procedure: Measuring the small instestine length using pre-marked laparoscopic graspers
- 3D CT scan group (Active Comparator): In this arm, all patients involved in the study will have a pre-operative CT scan, for which a 3D reconstruction will be done and measure the whole small intestinal length.
  Interventions: Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: CT — CT measurment of small bowel
  Arms: 3D CT scan group
Procedure: Measuring the small instestine length using pre-marked laparoscopic graspers — Intra-operatively, the surgeon will assess the length of the small intestine using a 5-cm marked laparoscopic graspers to accurately assess the whole small intestine length.
  Arms: Marked Laparoscopic graspers group

SUMMARY:
Measuring bowel length during hypo-absorptive surgeries like Roux-en-Y gastric bypass (RYGB) and Single Anastomosis Duodeno-ileal Sleeve (SADI-s) is controversial and usually abandoned due to the high risk of intestinal injury. However, some surgeons, especially in revisional surgery, prefer to count the whole bowel length to avoid leaving very short segments and severe malnutrition afterwards.

3D reconstructed CT scan can be useful in such conditions, avoiding the risk of intestinal injury, but accurate measures might be doubtful.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for revisional bariatric surgery
* Patients consenting to participate in the study.

Exclusion Criteria:

* Patients with severe adhesions where measuring the small bowel may expose them to unnecessary injuries.
* Patients refusing to participate in the study.
* Patient refusing CT scan to be done pre-operatively.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-26 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Accurate small bowel length | about 6 months
  the aim of the study to assess if the CT scan with 3D reconstruction will give accurate measures for the bowel length compared to the marked graspers used in laparoscopic surgery

SECONDARY OUTCOMES:
Operative time | intraoperative
  measuring the whole bowel length may increase the operative time according to the skills of the surgeon, the presence of adhesions, and short mesentery.
Intestinal Injury | up to 6 months
  counting the whole bowel length is a tedious procedure, especially in patients with obesity, where the mesentery is dense and may cause injury to the bowel.
  In this study, we will assess the incidence of intestinal injury of the small bowel, detected intra-operatively or post-operatively.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kasr Alainy Medical School, Cairo University, Cairo, Old Cairo
  - Kasr Alainy Medical School, Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Massalou D, Bege T, Bourgouin S, Mancini J, Masson C, Baque P, Berdah SV. Three-dimensional variability of the mesentery and the superior mesenteric artery: application to virtual trauma modeling. Surg Radiol Anat. 2014 May;36(4):401-8. doi: 10.1007/s00276-013-1178-1. Epub 2013 Jul 31. PMID 23900506
- [Background] Zorrilla-Nunez LF, Campbell A, Giambartolomei G, Lo Menzo E, Szomstein S, Rosenthal RJ. The importance of the biliopancreatic limb length in gastric bypass: A systematic review. Surg Obes Relat Dis. 2019 Jan;15(1):43-49. doi: 10.1016/j.soard.2018.10.013. Epub 2018 Oct 22. PMID 30501957
- [Background] Ahuja A, Tantia O, Goyal G, Chaudhuri T, Khanna S, Poddar A, Gupta S, Majumdar K. MGB-OAGB: Effect of Biliopancreatic Limb Length on Nutritional Deficiency, Weight Loss, and Comorbidity Resolution. Obes Surg. 2018 Nov;28(11):3439-3445. doi: 10.1007/s11695-018-3405-7. PMID 30032419
- [Background] Mahawar KK, Parmar C, Carr WRJ, Jennings N, Schroeder N, Small PK. Impact of biliopancreatic limb length on severe protein-calorie malnutrition requiring revisional surgery after one anastomosis (mini) gastric bypass. J Minim Access Surg. 2018 Jan-Mar;14(1):37-43. doi: 10.4103/jmas.JMAS_198_16. PMID 28695878
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12194548/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15376204/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/10022706/